CLINICAL TRIAL: NCT02327520
Title: The Burden of Clostridium Difficile Infection in Thai Population: the First Report in Southeast Asia by 2010 Nationwide Study
Brief Title: Clostridium Difficile Infection: the First Report in Southeast Asia by 2010 Nationwide Study
Status: Completed | Type: Observational
Sponsor: King Chulalongkorn Memorial Hospital (Other)
Responsible Party: Principal Investigator, Rapat Pittayanon, MD, Gastrointestinal Unit, King Chulalongkorn Memorial Hospital, King Chulalongkorn Memorial Hospital
Other Study IDs: RP009
Record Dates: First submitted 2014-12-22; First posted 2014-12-30 (Estimated); Last update posted 2014-12-30 (Estimated); Status verified 2014-12

CONDITIONS: Clostridium Difficile Infection
Keywords: Clostridium difficile infection; burden; nationwide study; South East Asia; Thailand; Epidemiology; Outcome Assessment (Health Care) [N04.761.559.590]
MeSH Terms: conditions — Clostridium Infections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Colitis with CDI: Patients who diagnosed with CDI will be analysed
  Interventions: Other: Colitis with CDI treatment

INTERVENTIONS:
Other: Colitis with CDI treatment — All patients will be treated with standard treatment

SUMMARY:
The authors retrieved in-patient medical data, including the expense, from the 2010 Thailand Nationwide Hospital Admission Database, which is part of the National Health Security Office (NHSO). The diagnosis of digestive diseases with any form of colitis listed in the causes, either as principal diagnosis or co-morbidity, coding by the ICD-10 was recorded. The inclusion criteria were: 1) diagnosis of enterocolitis due to Clostridium difficile (ICD10-A07); and 2) age of more than 18 years. If the data was incomplete, the case was excluded. The baseline characteristics, including age, sex, co-morbidity disease and history of endoscopy or surgery, were recorded. The burden of CDI was evaluated by length of hospital stay (LOS), mortality rate, and hospital charge.

ELIGIBILITY:
Inclusion Criteria:

* The patients with the diagnosis of Clostridium difficile (ICD10-A07)
* Age of more than 18 years.

Exclusion Criteria:

* Data incompleted

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients with the diagnosis of Clostridium difficile (ICD10-A07) with age of more than 18 years were included.
Sampling Method: Non-Probability Sample
Enrollment: 204666 (Actual)
Dates: Start 2010-01; Primary Completion 2010-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Death rate and length of hospital stay in CDI during admission | participants will be followed for the duration of hospital stay, an expected average of 2 weeks
  Length of hospital stay(LOS), mortality rate and hospital charge were used as the indicators for evaluating the burden of CDI.
Hospital charge of CDI | participants will be followed for the duration of hospital stay, an expected average of 2 weeks
  Length of hospital stay(LOS), mortality rate and hospital charge were used as the indicators for evaluating the burden of CDI.

CONTACTS AND LOCATIONS:
Overall Officials: Rapat Pittayanon, MD, Principal Investigator — King Chulalongkorn Memorial Hospital